CLINICAL TRIAL: NCT01298856
Title: The Effect of Hydrotherapy and Land-based Rehabilitation Program Combined With Ankle Taping on Ankle Functional Ability and Re-injury Rate in Athletes With Chronic Ankle Instability
Brief Title: The Effect of Hydrotherapy and Land-based Rehabilitation Program Combined With Ankle Taping in Athletes With Chronic Ankle Instability
Acronym: CAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Thammasat University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 014/52
Record Dates: First submitted 2011-01-08; First posted 2011-02-18 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-01

CONDITIONS: Sports Rehabilitation Program; Hydrotherapy; Ankle Instability
Keywords: hydrotherapy; chronic ankle instability; ankle taping
MeSH Terms: interventions — Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydrotherapy (Active Comparator): hydrotherapy and ankle taping and land based exercise
  Interventions: Procedure: hydrotherapy
- land-based (Active Comparator): land-based and ankle taping program
  Interventions: Procedure: hydrotherapy

INTERVENTIONS:
Procedure: hydrotherapy — hydrotherapy and ankle taping and land-based
  Other Names: ankle taping; land-based

SUMMARY:
There will be a difference in ankle functional ability between athletes with chronic ankle instability in the intervention group and in the control group.

ELIGIBILITY:
Inclusion Criteria:

* recurrent ankle sprain in one year
* sustain at least one repeated injury or have the experience of ankle instability feelings or "giving way"
* not undergoing formal or informal rehabilitation for the unstable ankle in the last three months
* have residual symptoms after recurrent sprain of the ankle

Exclusion Criteria:

* have the history of fracture or surgical procedures in the lower extremity
* have the history of neurological disorders affecting the lower extremities vestibular dysfunction or balance disorder
* allergic to the zinc oxide compound in the adhesive tape

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To compare the effect of ankle functional ability between the athletes with chronic ankle instability in the intervention group and the control group | 18 months

SECONDARY OUTCOMES:
To compare the effect of active joint position sense, single limb balance, SF-36 and re-injury rate | 18 months
  Parameters
  1. active joint position sense in ankle plantarflexion 30 degree and ankle inversion 15 degree
  2. single limb balance in standard deviation and Range
  3. SF-36 in 8 Items of questionnairs

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University, Khlong Luang, Changwat Pathum Thani, Thailand